CLINICAL TRIAL: NCT03955211
Title: A Phase 2 Open-Label Study of the Pharmacokinetics (PK) and Safety of HTX-011 Administered Postpartum to Women Undergoing a Planned Caesarean Section
Brief Title: HTX-011 Administration Study in Planned Caesarean Section Procedure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTX-011-220
Record Dates: First submitted 2019-05-09; First posted 2019-05-20 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Analgesia
Keywords: postoperative pain; caesarean section; C-section
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — KPNA1 protein, human; Ibuprofen; Acetaminophen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Treatment Group 1 (Experimental): A single dose of HTX-011 administered via instillation into the surgical site.
  Interventions: Drug: HTX-011; Device: Luer Lock Applicator
- Treatment Group 2 (Experimental): A single dose of HTX-011 administered via instillation into the surgical site and a scheduled non-opioid multimodal analgesic (MMA) regimen.
  Interventions: Drug: HTX-011; Device: Luer Lock Applicator; Drug: Ibuprofen; Drug: Acetaminophen

INTERVENTIONS:
Drug: HTX-011 — 300 mg
  Other Names: Cohort 1
  Arms: Treatment Group 1
Drug: HTX-011 — 400 mg
  Other Names: Cohort 2
  Arms: Treatment Group 2
Device: Luer Lock Applicator — Applicator for instillation.
Drug: Ibuprofen — 400 mg
  Arms: Treatment Group 2
Drug: Acetaminophen — 975 mg to 1 g
  Arms: Treatment Group 2

SUMMARY:
This is a Phase 2, open-label study to evaluate the PK and safety of HTX-011 in women undergoing a planned C-section.

ELIGIBILITY:
Inclusion Criteria:

* Is expected, at the time of Screening visit, to deliver a single neonate.
* Is scheduled to undergo a planned C-section surgery with a low transverse skin incision (eg, Pfannenstiel).
* Has American Society of Anesthesiologists (ASA) Physical Status of I, II, or III.
* Agrees to practice abstinence or use double-barrier contraception in the event of sexual activity and commits to the use of an acceptable form of birth control for 30 days after HTX-011 administration.
* Agrees to refrain from the use of breast milk from this pregnancy in any manner.

Exclusion Criteria:

* Has planned to breastfeed her neonate at any time during the 28-day period after HTX-011 administration.
* Has had a prior full-term pregnancy with unsuccessful breast milk expression.
* Has a planned concurrent surgical procedure.
* Has a contraindication or a known or suspected history of hypersensitivity or clinically significant idiosyncratic reaction to required study medications.
* Has been administered bupivacaine within 5 days prior to the scheduled surgery.
* Has been administered any local anesthetic within 72 hours prior to the scheduled surgery.
* Has been administered systemic steroids within 5 half-lives or 10 days prior to administration of study drug.
* Has initiated treatment with study medications within 1 month prior to study drug administration that can impact pain control.
* Has taken any NSAIDs within least 10 days prior to the scheduled surgery.
* Has current significant placental abnormality/complications including, but not limited to, placenta previa or placenta accreta.
* Has a medical condition such that, in the opinion of the Investigator, participating in the study would pose a health risk to the subject or confound the postoperative assessments.
* Has uncontrolled anxiety, psychiatric, or neurological disorder.
* Had a malignancy in the last year, with the exception of nonmetastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
* Has a known or suspected history of drug abuse, a positive drug screen on the day of surgery, or a recent history of alcohol abuse.
* Previously participated in an HTX-011 study.
* Received an investigational product or device in a clinical trial within 30 days or within 5 elimination half-lives.
* Weight is <50 kg at the time of Screening visit.
* In the Investigator's judgment, subject is likely to have been morbidly obese prior to her pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of bupivacaine, meloxicam, dimethyl sulfoxide (DMSO) and HTX-011 polymer | Day 1 to Day 16 for Cohort 1; Day 1 to Day 11 for Cohort 2
Time of maximum plasma concentration (Tmax) of bupivacaine, meloxicam, DMSO and HTX-011 polymer | Day 1 to Day 16 for Cohort 1; Day 1 to Day 11 for Cohort 2
Half life (t1/2) in plasma of bupivacaine, meloxicam, DMSO and HTX-011 polymer | Day 1 to Day 16 for Cohort 1; Day 1 to Day 11 for Cohort 2
Half life (t1/2) in milk of bupivacaine, meloxicam, DMSO and HTX-011 polymer | Day 1 to Day 16 for Cohort 1; Day 1 to Day 11 for Cohort 2
Amount of analyte excreted in breast milk over time (Ae) | Day 1 to Day 16 for Cohort 1; Day 1 to Day 11 for Cohort 2
Fraction of dose excreted in breast milk over time (Fe) | Day 1 to Day 16 for Cohort 1; Day 1 to Day 11 for Cohort 2

SECONDARY OUTCOMES:
Mean area under the curve of the NRS pain scores through 72 hours (AUC0-72). | 72 hours
Incidence of treatment-emergent adverse events (TEAEs). | 28 Days.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Helen Keller Hospital, Sheffield, Alabama
  - Sharp Mary Birch Hospital for Women and Newborns, San Diego, California
  - Duke University Medical Center, Durham, North Carolina
  - UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania